CLINICAL TRIAL: NCT02872805
Title: Adolescent to Adult Patient-centered HIV Transition (ADAPT) Study
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Vicki Tepper, Associate Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00070099
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEPFAR Enhanced Standard of Care (PESCA) (Active Comparator): This arm reflects an enhanced standard of care comparison group for PEPFAR supported sites. We will provide standardized materials to be used by current clinical staff to help support whatever the site specific activities are related to transition from pediatric to adult medical care
  Interventions: Other: PEPFAR Enhanced Standard of Care (PESCA)
- Peer Transition Advocate (PTA) (Experimental): The PTAs will be present during patient clinic appointments to mentor and support participants in the development of independent health care behaviors. They will engage patients in role-plays to simulate appointments in adult practices. The PTAs will accompany patients during the transition process to the adult providers, to inform, support, and facilitate their successful transition to adult care. PTA duties, performed in the clinic and in the community, will include psychosocial support; facilitation of disclosure; adherence counseling, monitoring, and support; screening of patients for significant signs of illness and referral for care; and tracking and defaulter tracing of patients. PTA will support counseling and testing services for adolescents within the facilities. For those perinatally-infected, important care and support services include disclosure and stigma issues.
  Interventions: Behavioral: Peer Transition Advocate (PTA)

INTERVENTIONS:
Other: PEPFAR Enhanced Standard of Care (PESCA) — Standardized materials will be provided to PEPFAR supported clinical sites to assist clinic teams with supporting patients in the transition from pediatric to adult medical care
  Other Names: Enhanced Standard of Care
  Arms: PEPFAR Enhanced Standard of Care (PESCA)
Behavioral: Peer Transition Advocate (PTA) — The PTAs will be present during patient clinic appointments to mentor and support participants in the development of independent health care behaviors. They will engage patients in role-plays to simulate appointments in adult practices. The PTAs will accompany patients during the transition process to the adult providers, to inform, support, and facilitate their successful transition to adult care. PTA duties, performed in the clinic and in the community, will include psychosocial support; facilitation of disclosure; adherence counseling, monitoring, and support; screening of patients for significant signs of illness and referral for care; and tracking and defaulter tracing of patients. PTA will support counseling and testing services for adolescents within the facilities. For those perinatally-infected, important care and support services include disclosure and stigma issues.
  Arms: Peer Transition Advocate (PTA)

SUMMARY:
One of the distinct challenges faced by emerging adults with HIV is the transition of their care from their long-term pediatric HIV provider to treatment within an adult HIV program. The consequences of an unsuccessful transition can range from difficult to catastrophic. The Adolescent to Adult Patient-centered HIV Transition (ADAPT) Study is a prospective cohort trial of an innovative intervention targeting gaps in care that are major drivers of loss in the ART continuum of care cascade among adolescents and increasing missed opportunities to engage adolescents into care.

DETAILED DESCRIPTION:
The specific aims of ADAPT are: 1. To inform strategies for transition services in resource-limited settings; 2. To examine the developmental, clinical, and other factors that predict a successful transition; and, 3. To gain fundamental insight on implementation barriers among African adolescents through the application of the ego-network defined social support that will inform targets for structured intervention. ADAPT will be conducted in central, southern, and northern Nigeria at selected PEPFAR sites supported by the Institute of Human Virology, Nigeria. To address Aim 1 the investigators will conduct six focus groups including: Adolescent patients, parents and health care providers. To address aim 2, the investigators will conduct a cluster randomized clinical trial. The two interventions are based on prior evidence-informed engagement strategies: 1) educational interventions and 2) interventions that use a peer transition advocate who prepares the adolescent and their parents for transition. The investigators will enroll 300 patients (150 patients in each arm). The sites will be assigned to either the intervention arm or a control arm. The primary outcome will be successful transition, keeping two follow-up appointments within a nine months period following transition. Secondary outcomes, as recommended by focus group participants will also be measured. To examine the potential role of social network components and characteristics of both egos and alters on primary outcomes, a Generalized Estimating Equation (GEE) approach will be used to explore the associations between primary outcomes and factors at the ego, alter, and network levels. The finding from this study will guide institution of best practices for transitioning adolescents in Nigeria and other countries lower and middle income countries with similar challenges and potential for high impact.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients between the ages of 16-19 years of age
* Patients who have been in care at the study site facility for a minimum of 1 year
* Patients who plan to transition their HIV care to one of the selected study sites
* Patients who are able to provide informed consent

Exclusion Criteria:

* HIV infected patients who have significant cognitive impairments(e.g., Mental retardation)
* Patients planning to transition their HIV care outside the selected study facilities

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 298 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Successful transition | 9 months after transition occurs
  ADAPT focuses on a service primary outcome, successful transition, which is defined as two consecutive kept appointments at the designated adult clinic within 9 months of transition
Viral load suppression | 12 months after transition occurs
  viral load (VL)<400 at 12 months post-transition

CONTACTS AND LOCATIONS:
Overall Officials: Vicki J Tepper, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Institute of Human Virology, Nigeria, Abuja, Federal Capital Territory, Nigeria

IPD SHARING:
Plan to Share IPD: No